CLINICAL TRIAL: NCT04283253
Title: Neurophysiological and Kinematic Predictors of Response in Chronic Stroke
Brief Title: Predictors of Response in Chronic Stroke
Acronym: SRT5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00003161
Record Dates: First submitted 2020-01-21; First posted 2020-02-25 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Stroke; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Stroke; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: One-arm, multiple baseline sequential, cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Robot + TTT Exercise (Experimental): All participants will be enrolled in this group to receive the same 60 minute study intervention consisting of wrist and shoulder-elbow robot training and TTT arm exercises.
  Interventions: Device: Robot + TTT exercise

INTERVENTIONS:
Device: Robot + TTT exercise — The intervention will be completed 36 visits approximately 3x/week for 12-18 weeks. The training progression will be sequential with 12 visits completed on the wrist robot, followed by 12 visits on the shoulder-elbow robot and completing with 12 visits alternating sessions on the wrist and shoulder-elbow robot. Participants will perform robot training for 45 minutes with each robot followed by 15 minutes of TTT practice to complete their 60 minute intervention session.

SUMMARY:
This study will validate a predictive model that uses demographics, functional status, neurophysiology, neuroanatomy, and other potential biomarkers to predict the likelihood of a clinically significant change in impairment at the end of a robot assisted therapy intervention.The study will include magnetic resonance imaging (MRI), transcranial magnetic stimulation (TMS), and an arm exercise program consisting of robot-assisted exercise combined with functional arm exercise called transition to task training (TTT).

DETAILED DESCRIPTION:
After informed consent, a baseline neurological exam, medical records review, MRI of the brain, TMS, questionnaires, cognitive testing, robot evaluations, and arm function testing will occur. Baseline testing will occur in the first 4-6 weeks of participation including two separate sessions approximately 1 week a part to examine arm strength, range of motion, and ability to perform functional tasks, with one additional session if needed to verify stability between results. Additionally, one robot evaluation will be completed.

The intervention phase consists of 12 weeks of robot and transition to task arm exercise training (TTT). Interventions will occur approximately 3 times per week for 12 weeks for a total of 36 visits. Additional time and visits will be allowed with visits occurring 4 times per week or up to 6 additional weeks (not to exceed 18 weeks) if scheduling conflicts arise. The intervention sessions will be one hour in duration.

During the hour-long intervention, 45 minutes of robotic intervention will be followed by 15 minutes of TTT. The training will be sequential with 12 sessions focused on the wrist, followed by 12 sessions on the shoulder-elbow and the final 12 sessions alternating between the wrist and elbow-shoulder.

After the final training session, subjects will return after a 12 week retention period. At various time points during and after the intervention phase there will be additional arm function testing, robot evaluations, questionnaires, MRI and TMS sessions for re-assessment.

ELIGIBILITY:
Inclusion Criteria:

* Clinically defined, unilateral, hemiparetic stroke with radiologic exclusion of other possible diagnosis
* Stroke onset at least 6 months before enrollment
* Present with Mild/Moderate to Severe arm dysfunction (based on Fugl-Meyer scores of 10 to 45)
* Be medically stable to participate in the study
* Be English speaking

Exclusion Criteria:

* Unable to give informed consent
* Have a serious complicating medical illness that would preclude participation.
* Contractures or orthopedic problems limiting range of joint motion in the potential study arm
* Visual loss such that the subject would not be able to see the test patterns on the robot computer monitor
* Botulinum toxin to study arm within four months of study enrollment or if received during the study period
* Unable to comply with requirements of the study
* Participants with a history of a seizure will not be precluded from the study, but will not be enrolled in the TMS portions
* Participants with electromagnetic exclusions (metal implants in the cranium, implanted electronic devices etc.) will not be precluded from the study but will be excluded from the MRI and TMS portions
* Have a serious complicating medical illness that would preclude participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Wittenberg, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared. Where practicable, sharing should take place under a written agreement prohibiting the recipient from identifying or re-identifying (or taking steps to identify or reidentify) any individual whose data are included in the dataset. However, it is permissible for final datasets in machine-readable format to be submitted to and accessed from PubMed Central (and similar sites) provided that care is taken to ensure that the individuals cannot be re-identified using other publicly available information.
  Datasets will be made available to the public following appropriate approvals for disclosure criteria.
  Every effort will be made to protect personal privacy and the confidentiality of private information collected for research purposes. This particular dataset will be de-identified and the minimum amount of information necessary to achieve the objectives of the research proposed will be collected and shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Mehrholz J, Pohl M, Platz T, Kugler J, Elsner B. Electromechanical and robot-assisted arm training for improving activities of daily living, arm function, and arm muscle strength after stroke. Cochrane Database Syst Rev. 2018 Sep 3;9(9):CD006876. doi: 10.1002/14651858.CD006876.pub5. PMID 30175845
- [Background] Stinear CM, Byblow WD, Ackerley SJ, Barber PA, Smith MC. Predicting Recovery Potential for Individual Stroke Patients Increases Rehabilitation Efficiency. Stroke. 2017 Apr;48(4):1011-1019. doi: 10.1161/STROKEAHA.116.015790. Epub 2017 Mar 9. PMID 28280137
- [Background] Connell LA, Smith MC, Byblow WD, Stinear CM. Implementing biomarkers to predict motor recovery after stroke. NeuroRehabilitation. 2018;43(1):41-50. doi: 10.3233/NRE-172395. PMID 30056436
- [Background] Lang CE, Bland MD, Bailey RR, Schaefer SY, Birkenmeier RL. Assessment of upper extremity impairment, function, and activity after stroke: foundations for clinical decision making. J Hand Ther. 2013 Apr-Jun;26(2):104-14;quiz 115. doi: 10.1016/j.jht.2012.06.005. Epub 2012 Sep 10. PMID 22975740
- [Background] Gauthier LV, Taub E, Mark VW, Perkins C, Uswatte G. Improvement after constraint-induced movement therapy is independent of infarct location in chronic stroke patients. Stroke. 2009 Jul;40(7):2468-72. doi: 10.1161/STROKEAHA.109.548347. Epub 2009 May 21. PMID 19461024

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Robot + TTT Exercise
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Robot + TTT Exercise
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: A Change in the Fugl-Meyer Upper Extremity Assessment Score
Description: The Fugl-Meyer is one of the primary outcome measures assessing change in arm use from baseline testing to mid-training after visits 12 and 24, and post-training after visit 36 and the 12 week retention period. It is a stroke-specific measure of impairment of the upper extremity that has been shown to be valid and reliable with high inter-rater and test-retest reliability. It provides a direct-observational assessment of volitional movement and motor impairment related to reflexes, sensation, and abnormal synergies. Each item on the FM is rated on a three-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully). The scale ranges from 0-66 with higher scores representing less motor impairment.
Time Frame: Immediately following the 12-week intervention
Population: Only one subject was enrolled and data collection was incomplete due to the Covid-19 pandemic. The evaluations following the 12-week intervention were not performed.
Measure: Number; unit: units on a scale
Arm/Group | Robot + TTT Exercise
Number analyzed (Participants) | 1
units on a scale
  Baseline One | 11
  Baseline Two | 12
  After Visit 12 | 13
  After Visit 24 | 14

2. Other Pre Specified Outcome: A Change in Motor Evoked Potential During Transcranial Magnetic Stimulation of the Motor Cortex
Description: TMS stimulation of the motor cortex will be performed using MagStim 200 Magnetic Stimulators (MagStim Ltd., Wales, UK) to assess change in the motor evoked potential (MEP) of the arm muscles.
Time Frame: Immediately following the 12-week intervention
Population: Only one subject was enrolled and data collection was incomplete due to the Covid-19 pandemic. The evaluations (including TMS) following the 12-week intervention were not performed.
Arm/Group | Robot + TTT Exercise
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: A Change in Brain Connections Assessed Via MRI of the Brain
Description: A detailed analysis of the MRI data will examine individual interregional connections to determine whether any of them are more sensitive to the intervention than others.
Time Frame: Immediately following the 12-week intervention
Population: MRI was not collected as the one enrolled subject did not pass the MRI safety screening.
Arm/Group | Robot + TTT Exercise
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Robot + TTT Exercise
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT04283253/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT04283253/ICF_001.pdf